CLINICAL TRIAL: NCT00305955
Title: Bilateral Refractive Amblyopia Treatment Study
Acronym: ATS7
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Director, Jaeb Center for Health Research
Other Study IDs: NEI-101; 2U10EY011751 (NIH)
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-10

CONDITIONS: Bilateral Refractive Amblyopia
Keywords: amblyopia; bilateral amblyopia; refractive error
MeSH Terms: conditions — Amblyopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spectacles — optimal spectacle correction

SUMMARY:
The purpose of this study will be to:

* Determine the amount of visual acuity improvement with treatment of presumed bilateral refractive amblyopia
* Determine the time course of visual acuity improvement with treatment

DETAILED DESCRIPTION:
There is a paucity of literature on bilateral amblyopia that is due to a substantial amount of refractive error (hypermetropia or astigmatism), and it is limited principally to review articles and case reports. The incidence is not known, but in one study, 4 of 830 (0.5%) children examined at the time of entry into school had bilateral amblyopia. Schoenleber et al performed a retrospective review of office records and identified 184 children with > +4.00 diopters of hypermetropia in both eyes, 12 of whom (6.5%) had bilateral amblyopia of 20/50 or worse. Ten of the 12 children (83%) improved to 20/40 or better in both eyes over a mean follow-up time of 22 months. Werner and Scott reported 6 cases of bilateral hypermetropic amblyopia with a spherical equivalent of at least +5.00 D and an initial visual acuity of 20/40 or worse in both eyes. All 5 patients with follow up improved with glasses alone, and 2 of these 5 had a most recent visual acuity worse than 20/40 in one eye with follow-up less than one year. Cavazos et al identified 218 eyes with hyperopia > +5.00 D or astigmatism >+2.00 D. Of these, 82 (38%) of the dominant eyes had an initial corrected visual acuity less than 20/25. Most improved to > 20/25, but many patients were lost to follow-up. In ongoing studies, bilateral refractive amblyopia is being evaluated in Native Americans.

1. Patients will be enrolled who have bilateral refractive error with hyperopia >+4.00 D and/or astigmatism >2.00 D and have visual acuity in each eye, measured using best correction derived from cycloplegic refraction, meeting the following criteria:

   * Using E-ETDRS testing for patients age 7 to <11 years: visual acuity 20 to 70 letters (20/40 to 20/400)
   * Using ATS HOTV testing for patients age 3 to <7 years visual acuity 20/50 to 20/400
2. Enrolled patients will be prescribed spectacles, which will be paid for by the study.
3. The patient will return for a Spectacle Baseline visit within 30 days, at which time the spectacles will be placed on the patient for the first time and binocular and monocular visual acuities will be measured.

   * Patients whose monocular acuity at the Spectacle Baseline Visit is 20/25 or better in both eyes will end the study
   * Patients whose monocular acuity at the Spectacle Baseline Visit is worse than 20/25 in at least one eye will begin a one-year period of study follow up
4. Follow-up visits are required at 5±:1 week, 13±:2 weeks, 26±:4 weeks, and 52±:4 weeks.

   * If at any follow-up visit a patient's monocular acuity is 20/25 or better in both eyes, the patient should return for the 52-week visit only and may skip the interim follow-up visits.

Sample size: The study plans to enroll 100 patients. At least 50 patients will be enrolled who have an interocular difference of less than 3 lines by ATS HOTV or less than 15 letters by E-ETDRS at the Spectacle Baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to <11 years
* Able to perform single-surrounded single optotype visual acuity using the ATS HOTV protocol for children 3 to <7 years old and using the E-ETDRS protocol for children 7 to <11 years old
* Monocular visual acuity in each eye, measured using trial frames or phoropter with best correction derived from cycloplegic refraction, meeting the following criteria:
* Using E-ETDRS testing for patients age 7 to <11 years: visual acuity 20 to 70 letters (20/40 to 20/400)
* Using ATS HOTV testing for patients age 3 to <7 years acuity 20/50 to 20/400
* Refractive error that meets at least one of the following criteria in each eye:
* Spherical equivalent >+4.00 D
* Astigmatism >2.00 D
* Investigator believes that the patient's reduced visual acuity is due to bilateral, refractive amblyopia
* Investigator not planning to prescribe occlusion, patching or any other amblyopia treatment other than spectacles at this time
* Cycloplegic refraction and ocular examination within 2 months prior to enrollment

Exclusion Criteria:

* Myopia greater than -6.00 D of spherical power in plus cylinder form
* Ocular cause for decreased acuity in either eye; nystagmus per se will not exclude a patient from the study
* Refractive correction (spectacles or contact lenses) in past three months and no more than one month of refractive correction ever
* Prior treatment for amblyopia (other than the refractive correction permitted in previous exclusion criteria)
* Prior intraocular or refractive surgery
* Use of contact lenses during the study

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Visual acuity of 20/25 or better in both eyes | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David K. Wallace, M.D., Principal Investigator — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Wallace DK, Chandler DL, Beck RW, Arnold RW, Bacal DA, Birch EE, Felius J, Frazier M, Holmes JM, Hoover D, Klimek DA, Lorenzana I, Quinn GE, Repka MX, Suh DW, Tamkins S; Pediatric Eye Disease Investigator Group. Treatment of bilateral refractive amblyopia in children three to less than 10 years of age. Am J Ophthalmol. 2007 Oct;144(4):487-96. doi: 10.1016/j.ajo.2007.05.040. Epub 2007 Aug 20. PMID 17707330